CLINICAL TRIAL: NCT03704961
Title: Professor (Head of the Departmant of Nursing)
Brief Title: Effect of Auditory Distractions on Pediatric Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, nurcan özyazıcıoğlu, UludagU, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- classical music (Experimental)
  Interventions: Behavioral: music and audiobook listening
- Turkish music (Experimental)
  Interventions: Behavioral: music and audiobook listening
- audiobook (Experimental)
  Interventions: Behavioral: music and audiobook listening

INTERVENTIONS:
Behavioral: music and audiobook listening

SUMMARY:
The aim of the study was to determine the effect of different auditorial methods of attention distraction on postoperative pain and anxiety in children. Three group pre and post-test randomized clinical trial.The data were collected using the Socio-demographic Data Form for Child and Parent, Visual Analogue Scale, Wong-Baker Faces Pain Scale and State-Trait Anxiety Inventory for Children. The investigators found that listening to classical music, Turkish music and audiobook methods played an effective role in decreasing postoperative pain and anxiety state in children in the three groups in the study. As a result, investigators showed that different auditorial attention distraction methods had a decreasing effect on postoperative pain and anxiety in children.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 7-14 years old,
* staying in a single room,
* those for whom a surgical procedure for inguinal or abdominal region had been planned,
* in the first hour of postoperative period,
* free of any problem that prevents expression of the post-operative pain,
* free of hearing problems,
* having undergone same analgesia protocol; were included in the study.

Exclusion Criteria:

-

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | one hour after the patients were taken to the patient's room after the surgery
  Visual Analog Scale (VAS): It is a straight line with a length of 10 cm. On the '0 line', there is "no pain" and on the '10 line', it is "unbearable pain". The child is asked to mark the place indicating the severity of his/her pain.
Wong-Baker Faces Pain Scale | one hour after the patients were taken to the patient's room after the surgery
  This was developed by Donna Lee Wong and Connie Morain Baker. This scale is used to determine the level of pain in children over three years of age. The severity of pain is determined by the child with choosing the face that describes the child's pain level on the scale starting with the smiling face and ending with the crying face.
State-Trait Anxiety Inventory for Children | one hour after the patients were taken to the patient's room after the surgery
  This was developed by Spielberger (1973). It is a three-point Likert-type scale. The validity and reliability of the scale were performed by Özusta (1993).The scale consists of two parts as; 'state anxiety scale' and 'trait anxiety scale'. It consists of 40 items in total, 20 items in each part. The STAI-C was adapted from an adult scale and is also known as the "How I Feel Questionnaire". ıt comprises separate self-report scales for measuring two distinct anxiety concepts: state anxiety (S-Anxiety) and trait anxiety (T- Anxiety). The 20- item scale asseses a number of symptoms of anxiety such as "I get a funny feeling in my stomach" and "I am checking one of three alternatives that describes him or her best or indicates frequency of occurrence ( 1 = almost never; 2 = sometimes; 3 = often ).

SECONDARY OUTCOMES:
Visual Analogue Scale | Immediately after the listening was over
  Visual Analog Scale (VAS): It is a straight line with a length of 10 cm. On the '0 line', there is "no pain" and on the '10 line', it is "unbearable pain". The child is asked to mark the place indicating the severity of his/her pain.
Wong-Baker Faces Pain Scale | Immediately after the listening was over
  This was developed by Donna Lee Wong and Connie Morain Baker. This scale is used to determine the level of pain in children over three years of age. The severity of pain is determined by the child with choosing the face that describes the child's pain level on the scale starting with the smiling face and ending with the crying face.
State-Trait Anxiety Inventory for Children | Immediately after the listening was over
  This was developed by Spielberger (1973). It is a three-point Likert-type scale. The validity and reliability of the scale were performed by Özusta (1993).The scale consists of two parts as; 'state anxiety scale' and 'trait anxiety scale'. It consists of 40 items in total, 20 items in each part. The STAI-C was adapted from an adult scale and is also known as the "How I Feel Questionnaire". ıt comprises separate self-report scales for measuring two distinct anxiety concepts: state anxiety (S-Anxiety) and trait anxiety (T- Anxiety). The 20- item scale asseses a number of symptoms of anxiety such as "I get a funny feeling in my stomach" and "I am checking one of three alternatives that describes him or her best or indicates frequency of occurrence ( 1 = almost never; 2 = sometimes; 3 = often ).

IPD SHARING:
Plan to Share IPD: No